CLINICAL TRIAL: NCT04460703
Title: Persuasive Messages for COVID-19 Vaccine Uptake: a Randomized Controlled Trial, Part 1
Brief Title: COVID-19 Vaccine Messaging, Part 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000027983
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Vaccination; COVID-19
Keywords: messaging
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: In this study, 2/15 of participants will be assigned to a control message (bird feeding passage), 3/15 of sample to a baseline vaccine message, and 1/15 to each of the 10 other treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Control (Sham Comparator): Control message about birdfeeding
  Interventions: Other: Control message
- Baseline message (Active Comparator): These participants will be assigned a message about the benefits of vaccination. All other treatment arms include this baseline language.
  Interventions: Other: Baseline message
- Personal freedom (Experimental): Experimental message arm.
  Interventions: Other: Personal freedom message
- Economic freedom (Experimental): Experimental message arm.
  Interventions: Other: Economic freedom message
- Social benefit, self-interest (Experimental): Experimental message arm.
  Interventions: Other: Self-interest message
- Social benefit, community interest (Experimental): Experimental message arm.
  Interventions: Other: Community interest message
- Economic benefit (Experimental): Experimental message arm.
  Interventions: Other: Economic benefit message
- Social pressure- guilt (Experimental): Experimental message arm.
  Interventions: Other: Guilt message
- Social pressure- embarrassment (Experimental): Experimental message arm.
  Interventions: Other: Embarrassment message
- Social pressure- anger (Experimental): Experimental message arm.
  Interventions: Other: Anger message
- Trust in science (Experimental): Experimental message arm.
  Interventions: Other: Trust in science message
- Not bravery arm (Experimental): Experimental message arm.
  Interventions: Other: Not bravery message

INTERVENTIONS:
Other: Control message — 2/15 of the sample will be assigned to the pure control group, which is a passage on the costs and benefits of bird feeding.
  Arms: Control
Other: Baseline message — 3/15 of the sample will be assigned to a control group with a message about the effectiveness and safety of vaccines.
  Arms: Baseline message
Other: Personal freedom message — 1/15 of the sample will be assigned to this intervention, which is a message about how COVID-19 is limiting people's personal freedom and by working together to get enough people vaccinated society can preserve its personal freedom.
  Arms: Personal freedom
Other: Economic freedom message — 1/15 of the sample will be assigned to this intervention, which is a message about how COVID-19 is limiting peoples's economic freedom and by working together to get enough people vaccinated society can preserve its economic freedom.
  Arms: Economic freedom
Other: Self-interest message — 1/15 of the sample will be assigned to this intervention, which is a message that COVID-19 presents a real danger to one's health, even if one is young and healthy. Getting vaccinated against COVID-19 is the best way to prevent oneself from getting sick.
  Arms: Social benefit, self-interest
Other: Community interest message — 1/15 of the sample will be assigned to this intervention, which is a message about the dangers of COVID-19 to the health of loved ones. The more people who get vaccinated against COVID-19, the lower the risk that one's loved ones will get sick. Society must work together and all get vaccinated.
  Arms: Social benefit, community interest
Other: Economic benefit message — 1/15 of the sample will be assigned to this group, which is a message about how COVID-19 is wreaking havoc on the economy and the only way to strengthen the economy is to work together to get enough people vaccinated.
  Arms: Economic benefit
Other: Guilt message — 1/15 of the sample will be assigned to this message. The message is about the danger that COVID-19 presents to the health of one's family and community. The best way to protect them is by getting vaccinated and society must work together to get enough people vaccinated. Then it asks the participant to imagine the guilt they will feel if they don't get vaccinated and spread the disease.
  Arms: Social pressure- guilt
Other: Embarrassment message — 1/15 of the sample will be assigned to this message. The message is about the danger that COVID-19 presents to the health of one's family and community. The best way to protect them is by getting vaccinated and by working together to make sure that enough people get vaccinated. Then it asks the participant to imagine the embarrassment they will feel if they don't get vaccinated and spread the disease.
  Arms: Social pressure- embarrassment
Other: Anger message — 1/15 of the sample will be assigned to this message. The message is about the danger that COVID-19 presents to the health of one's family and community. The best way to protect them is by getting vaccinated and by working together to make sure that enough people get vaccinated. Then it asks the participant to imagine the anger they will feel if they don't get vaccinated and spread the disease.
  Arms: Social pressure- anger
Other: Trust in science message — 1/15 of the sample will be assigned to this message about how getting vaccinated against COVID-19 is the most effective way of protecting one's community. Vaccination is backed by science. If one doesn't get vaccinated that means that one doesn't understand how infections are spread or who ignores science.
  Arms: Trust in science
Other: Not bravery message — 1/15 of the sample will be assigned to this message which describes how firefighters, doctors, and front line medical workers are brave. Those who choose not to get vaccinated against COVID-19 are not brave.
  Arms: Not bravery arm

SUMMARY:
This study tests different messages about vaccinating against COVID-19 once the vaccine becomes available. Participants are randomized to 1 of 12 arms, with one control arm and one baseline arm. We will compare the reported willingness to get a COVID-19 vaccine at 3 and 6 months of it becoming available between the 10 intervention arms to the 2 control arms.

Study participants are recruited online by Lucid, which matches census based sampling in online recruitment.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* US resident

Exclusion Criteria:

* Younger than 18 years of age
* Non-US resident
* Do not consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Intention to get COVID-19 vaccine | Immediately after intervention, in the same survey in which the intervention message is provided
  This is a self reported measure, immediately after the intervention message, of the likelihood of getting a COVID-19 vaccination within 3 months and then 6 months of it becoming available. During analysis, responses among those assigned to different intervention messages will be compared to those in the control group.

SECONDARY OUTCOMES:
Vaccine confidence scale | Immediately after intervention, in the same survey in which the intervention message is provided
  This is a validated scale. This scale will be used to assess the impact of the messages on vaccine confidence. (Outcome assessed only for the half of the sample that answers these items post-treatment)
Persuade others item | Immediately after intervention, in the same survey in which the intervention message is provided
  This is a measure of a willingness to persuade others to take the COVID-19 vaccine.
Fear of those who have not been vaccinated | Immediately after intervention, in the same survey in which the intervention message is provided
  This is a measure of a comfort with an unvaccinated individual visiting an elderly friend after a vaccine becomes available
Social judgment of those who do not vaccinate | Immediately after intervention, in the same survey in which the intervention message is provided
  This is a scale composed of 4 items measuring the trustworthiness, selfishness, likeableness, and competence of those who choose not to get vaccinated after a vaccine becomes available

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data and analysis code will be posted in a public replication archive after publication.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After publication
Access Criteria: Anonymized data and analysis code will be posted in a public replication archive

REFERENCES:
- [Result] James EK, Bokemper SE, Gerber AS, Omer SB, Huber GA. Persuasive messaging to increase COVID-19 vaccine uptake intentions. Vaccine. 2021 Dec 3;39(49):7158-7165. doi: 10.1016/j.vaccine.2021.10.039. Epub 2021 Oct 22. PMID 34774363